CLINICAL TRIAL: NCT06680193
Title: Daily Affect and Cognition Impacts of Processing of Positive Memories Technique (PPMT) in a Trauma-Exposed Community Sample
Brief Title: Therapeutic Effects of the Processing of Positive Memories Technique on Posttrauma Health
Acronym: PPMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas, Denton, TX (Other)
Collaborators: University of Haifa, Israel (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-21-420; 2020017 (Other Grant/Funding Number: United States-Israel Binational Science Foundation)
Record Dates: First submitted 2024-10-30; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-10

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Posttrauma Health; Positive Autobiographical Memories; Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Processing of Positive Memories Technique (Experimental): PPMT was administered as a 4-session protocol in this arm.
  Interventions: Behavioral: Processing of Positive Memories Technique

INTERVENTIONS:
Behavioral: Processing of Positive Memories Technique — PPMT was administered weekly as a 4-session protocol. In session 1, participants receive psychoeducation on PTSD symptoms, an overview of PPMT, and are assessed for psychological symptoms. Sessions 1-4 involve the detailed processing of a salient positive autobiographical memory to elicit "values, affect, strengths, and thoughts" related to that positive memory. Homework assignments include listening to an audio recording of that memory, completing a "values, affect, strengths, and thoughts" log, and engaging in a behavioral activity. In session 4, the therapist also reviews psychological symptoms and addresses termination.

SUMMARY:
The current study will examine daily-level impacts of a technique addressing positive memory retrieval on thoughts, feelings, and health among individuals with trauma experiences.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is primarily a memory encoding- and retrieval-based disorder. If untreated, there are significant physical, psychological, social, and economic impacts for an individual, their families, and the society broadly. Research demonstrates that positive memory processes contribute to the etiology and maintenance of PTSD symptoms. Indeed, difficulties in retrieving and discussing positive memories are amplified among individuals with PTSD. Further, interventions capitalizing on (positive) memory retrieval have been linked to enhanced psychological well-being.

Considering this literature, the Processing of Positive Memories Technique (PPMT) was developed as a promising new treatment approach for posttraumatic stress disorder (PTSD), which involves detailed narration and processing of specific positive autobiographical memories. This study uses an innovative research protocol that combines case-series design and daily diary approaches to the effects of PPMT on daily affect, daily cognitions, and daily PTSD symptoms. It is hypothesized that at the daily level, in comparison to their an individual's pre-PPMT levels, following the PPMT intervention, participants will report (1) a lower count of endorsed daily PTSD symptoms, (2) increases in daily positive affect and decreases in daily negative affect, (3) increases in positive affect reactivity to daily positive events, and (4) decreases in daily posttrauma cognitions.

ELIGIBILITY:
Inclusion Criteria:

* being aged between 18 and 65 years
* endorsing a trauma with posttrauma symptoms
* access to an electronic device with internet capabilities
* working knowledge of English
* being a current resident of the Dallas Fort Worth metroplex
* willingness and availability to participate in approximately 10 weeks of this study (including 4 therapy sessions)
* willingness to be video-recorded during sessions for quality control purposes

Exclusion Criteria:

* active suicidal plan, suicidal attempt, homicidal plan, or homicidal attempt (past 3 months including current)
* currently in therapy with a mental health provider

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Daily negative and positive affect levels | Each day for 21 days prior to and after the intervention and each survey references the past 24 hours
  Daily Positive and Negative Affect are assessed by rating the extent of four positive (excited, cheerful, satisfied, relaxed) and six negative (stressed, irritated, anxious, sad, hopeless, insecure) emotions. This is adapted from the 20-item Positive and Negative Affect Scale. The total positive affect subscale score can range from 1 to 20, with higher scores reflecting more positive affect levels. The total negative affect subscale score can range from 1 to 30, with higher scores reflecting more negative affect.
Daily positive events | Each day for 21 days prior to and after the intervention and each survey references the past 24 hours
  Daily positive events is measured by 1 item which asked participants to think about the most positive event of the day and rate how pleasant it was. The score can range from 1 to 4, with higher scores reflecting that the event was more pleasant.
Daily posttrauma cognitions | Each day for 21 days prior to and after the intervention and each survey references the past 24 hours
  A 9-item brief version of the Posttraumatic Cognitions Inventory (PTCI-9) will measure trauma-related thoughts/beliefs with the time frame modified to 'in the last 24 hours.' The total raw score can range from 1 to 63, with higher scores reflecting endorsement of more negative posttrauma cognitions.
Daily PTSD symptoms | Each day for 21 days prior to and after the intervention and each survey references the past 24 hours
  Daily-life version of the Primary Care-PTSD-5 screen (PC-PTSD-5) will assess daily PTSD symptoms with the time frame modified to 'in the last 24 hours.' The total score can range from 0 to 5, with higher scores reflecting endorsement of more PTSD symptoms.
Number of retrieved positive memories | Baseline survey approximately 4 weeks prior to the intervention
  AMT assesses the number of retrieved positive memories by using five cue words followed by a prompt to recall a personally meaningful and specific memory of an event that took place within any 24-hour period. The total score could range from 0 to 5, with higher scores indicating more number of retrieved positive memories.
Number of retrieved positive memories | 1 week after intervention sessions
  AMT assesses the number of retrieved positive memories by using five cue words followed by a prompt to recall a personally meaningful and specific memory of an event that took place within any 24-hour period. The total score could range from 0 to 5, with higher scores indicating more number of retrieved positive memories.

SECONDARY OUTCOMES:
Positive Emotion Dysregulation | Baseline survey approximately 4 weeks prior to the intervention
  The Difficulties in Emotional Regulation Scale-Positive Emotions is a 13-item self-report measure that examines dysregulation of positive emotions. The total score could range from 1 to 65, with higher scores indicating more positive emotion dysregulation.
Positive Emotion Dysregulation | 1 week after intervention sessions
  The Difficulties in Emotional Regulation Scale-Positive Emotions is a 13-item self-report measure that examines dysregulation of positive emotions. The total score could range from 1 to 65, with higher scores indicating more positive emotion dysregulation.
Positive Emotion Dysregulation | At each of the 4 weekly intervention sessions and each survey references the past week
  The Difficulties in Emotional Regulation Scale-Positive Emotions is a 13-item self-report measure that examines dysregulation of positive emotions. The total score could range from 1 to 65, with higher scores indicating more positive emotion dysregulation.
PTSD symptom severity | Baseline survey approximately 4 weeks prior to the intervention
  The PTSD Checklist for DSM-5 is a 20-item self-report measure that will be used to evaluate PTSD symptom severity in relation to the worst trauma. The total score could range from 0 to 80, with higher scores reflecting more PTSD symptom severity.
PTSD symptom severity | 1 week after intervention sessions
  The PTSD Checklist for DSM-5 is a 20-item self-report measure that will be used to evaluate PTSD symptom severity in relation to the worst trauma. The total score could range from 0 to 80, with higher scores reflecting more PTSD symptom severity.
PTSD symptom severity | At each of the 4 weekly intervention sessions and each survey references the past week
  The PTSD Checklist for DSM-5 is a 20-item self-report measure that will be used to evaluate PTSD symptom severity in relation to the worst trauma. The total score could range from 0 to 80, with higher scores reflecting more PTSD symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Texas, Denton, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: De-identified IPD will be shared in 2029 until 2034.
Access Criteria: De-identified IPD will be stored with limited access in a data repository. Any interested researchers will email the PIs and complete a data sharing contract. If the contract is approved by the PIs, data will be shared in a secure manner.

REFERENCES:
- [Background] Greene T, Contractor AA, Dicker-Oren SD, Fentem A, Sznitman SR. The Effects of the Processing of Positive Memories Technique on Posttrauma Affect and Cognitions Among Survivors of Trauma: Protocol for a Daily Diary Study. JMIR Res Protoc. 2024 Jan 12;13:e51838. doi: 10.2196/51838. PMID 38214953
- [Derived] Rodenbaugh MM, Thompson LM, Sznitman SR, Jin L, Contractor AA. Refining processing of positive memories technique: client perspectives on components, format, and feasibility. Eur J Psychotraumatol. 2025 Dec;16(1):2563197. doi: 10.1080/20008066.2025.2563197. Epub 2025 Oct 9. PMID 41065062